CLINICAL TRIAL: NCT04266223
Title: Surface Monitoring Technology to Remove The Mask - Stage 1
Acronym: SMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: Western Sydney Local Health District (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SMART; U1111-1248-2457 (Registry Identifier: WHO UTN)
Record Dates: First submitted 2019-12-09; First posted 2020-02-12 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Head and Neck Cancer; Radiation Therapy Complication; Anxiety
Keywords: Radiation Therapy; Mask; Anxiety; Motion sickness; Claustrophobia
MeSH Terms: conditions — Head and Neck Neoplasms; Anxiety Disorders; Motion Sickness; Claustrophobia

STUDY DESIGN:
Intervention Model Description: This is a hypothesis-producing feasibility study that does not involve power calculations. The number of participants (20) was chosen to enable confidence in the primary outcome calculation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mask-free surface monitoring (Experimental): Lay in treatment position for 20 minutes with surface monitoring technology activated
  Interventions: Device: Mask-free surface monitoring

INTERVENTIONS:
Device: Mask-free surface monitoring — Mask-free headrest and couch for patient positioning for radiation therapy combined with a surface monitoring system

SUMMARY:
A pilot-stage device feasibility study investigating a mask-free motion-monitoring patient immobilisation system for use during radiation therapy treatment of head and neck cancer (HNC). This mask-free system combines the standard radiation therapy (RT) head rest to help the patient remain still with a surface guidance detection system that uses sensors to detect and track patient movement.

Patients who will have RT treatment for head and neck cancer involving an immobilisation mask will be asked to lie on the treatment couch for the normal treatment fraction time while the surface monitoring system is activated. We will then assess:

i) The level of acceptance of the system by HNC patients currently being treated with RT using an immobilisation mask, and ii) The ability of the surface guidance system to monitor movement of the patients

DETAILED DESCRIPTION:
Radiation therapy (RT) is a central treatment modality for 74% of head and neck cancer (HNC) patients where preservation of the form and function of localised organs and tissue is of prime importance. Radiation therapy offers the possibility of organ preservation by providing a non-surgical approach to curative treatment, while helping to limit the extent of surgery in cases where definitive surgery is unavoidable. Radiation therapy also has an important role in maintaining quality of life in the palliative management of incurable HNC, where it can prevent and alleviate pain, bleeding, tumour fungation and difficulty with swallowing, breathing and speech.

State-of-the-art RT for HNC delivers lethal radiation doses to the cancer while sparing vital organs situated just a few millimetres away. To achieve this level of accuracy, tight-fitting thermoplastic head and neck masks are used to immobilise the patient in the desired treatment position for the duration of each of their RT treatments. These thermoplastic immobilisation devices are accepted internationally as the necessary standard and included in published guidelines. Open masks are an emerging immobilisation measure and a first step to reduce patient discomfort and anxiety. An open mask has a smaller visual restriction and fewer restraint points.

Although, thermoplastic immobilisation masks are the accepted clinical standard for HNC RT, it is widely recognised and acknowledged that there are several limitations with their use. Changes to the mask's fit may be needed due to patient weight loss, tumour shrinkage, or treatment related oedema. Thus, radiation therapists are required to monitor the mask for fit throughout the treatment course, undertake imaging at regular intervals and make corrections as per published guidelines and local protocols. There is also risk of movement of the patient within the mask, which may lead to under dosing of the target and overdosing of organs at risk. Court et al. reported that patients in their study needed to be repositioned in the immobilisation mask before treatment for 14% of fractions; 30% of the repositioning was for shoulder shifts of 1 cm or greater. Neubauer et al. observed shoulder motion of 2-5 mm in each direction on average (20 mm max). These shifts resulted in coverage loss (dose to 99% of the clinical target volume decreased by up to 1Gy) or increased dose to organs at risk (e.g., dose to brachial plexus increased by 0.7Gy).

The ACRF Image X Institute at the University of Sydney has developed a novel surface guidance system that can be mounted to any RT imaging and treatment couch. This system is currently being used in a clinical trial (NCT02881203) to guide breast cancer patients into a reproducible breath hold: the patient's chest position is measured via surface imaging and the system delivers visual feedback to the patient via a screen for the patient to correct their breath hold level if necessary (i.e., surface guidance). This system uses off-the-shelf electronics, most importantly a sensor which includes an optical and a depth camera, delivering frames at a rate of 30Hz and allowing the patient and operator to see an augmented reality video feed, including the surface depth information.

Similar to this, we will apply optical and depth cameras for head and neck surface monitoring by integrating a second sensor and adapting it to the different location of treatment

Pilot-stage, single-arm study investigating the technical feasibility and patient acceptance of a non-interventional, non-invasive, mask-free surface detection system.

Towards the end of their scheduled radiation therapy treatments, people being treated for HNC with RT using a thermoplastic immobilisation mask will be asked to lie in a treatment position on a treatment couch using a standard radiation therapy headrest without the mask, for the normal amount of time taken for individual radiation therapy treatments (20 minutes). During this time, the mask-free surface detection system will detect and record their location and movement. Data collected by the surface detection system during this couch session will be analysed to determine the feasibility of using the equipment to detect location and movement over this period. Data collected directly from the participants immediately before, during and following the couch session will be used to determine their acceptance of the system in terms of comfort and anxiety when compared with wearing the mask, and any suggestions for improvement of the system. Data collected directly from the radiation therapists following the couch session will be used to investigate their thoughts on the abilities of the system, ease of use and suggestions they may have.

To investigate the effect of changes in appearance due to weight loss over the course of HNC radiation therapy treatment, a 5-minute surface monitoring couch session conducted before the start of radiation therapy will record baseline surface-monitoring information only.

Data analysis will occur at the University of Sydney outside of participant sessions.

ELIGIBILITY:
Inclusion Criteria

* A diagnosis of head and neck cancer, any stage
* ≥ 18 years of age
* ECOG performance status 0-2
* Receiving radiation therapy for HNC with a thermoplastic immobilisation mask
* Any other prior therapy allowed
* Willing and able to comply with all study requirements
* Must be able to read and complete questionnaires in English

Exclusion Criteria

* People with cognitive impairment which would preclude them from providing informed consent
* People who are unable to speak and read English and for whom obtaining consent would be difficult.

Withdrawal Criteria

* Participants may withdraw from the study at any time before, during or after participation, and do not have to provide a reason. They may do so by advising any member of the study team, research office or their treating team, by completing the withdrawal of consent form, verbally or in writing.
* Participants may be withdrawn from the study by the principal investigator, treating physician or attending clinician if they perceive the participant is experiencing or will likely experience physical or mental harm
* No additional study data will be collected for a participant after they withdraw from the study
* Withdrawing participants' data will be used unless the participant specifies they no longer give permission for the data to be stored or used, however, their data will not be removed from any analysis or publication that has already occurred, or from study databases once it has been de-identified
* Participant will be replaced if they withdraw or are withdrawn from the study prior to starting the second couch session. This will be done by recruitment of an additional participant.
* If a couch session is ended by the researcher or participant for reasons unrelated to the study (e.g. not related to equipment failure or participant non-acceptance), the session may be rescheduled, or participant replaced.
* Reasons for withdrawal will be reported in any outcome publications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Continuous acquisition of position and motion data of anatomical structures by the surface monitoring system | 20 minutes
  Technical feasibility of surface-monitoring system in ≥90% of consumers - operates continuously throughout the session and provides information on the position and motion of the cranium, mandible and shoulders without obvious erroneous results or faults
Patient acceptance of the surface monitoring system | 10 minutes
  Patients complete the session AND give a mean score of 4 or more for both comfort and acceptability on a Likert scale of 1-7, where 1 = 'Very Strongly Disagree' and 7 = 'Very Strongly Agree'

SECONDARY OUTCOMES:
Patient experience | 45 minutes
  Qualitative semi-structured interview of patient experience of interacting with the surface monitoring system and how that compared with the experience of the immobilisation mask during their radiation therapy treatment.
Radiation therapists' experience | 5 minutes
  Questionnaire of radiation therapist's experience scored according to a Likert scale of 1-5 where 1 = 'Strongly Disagree' and 5 = 'Strongly Agree'
Absolute Residual Motion of cranial and upper torso anatomy | 20 minutes
  Distance and direction of, and correlation between, motion of the cranial and upper torso anatomy relative to the fixed isocentre
Relative Residual Motion of cranial and upper torso anatomy | 20 minutes
  Distance and direction of, and correlation between, motion of the cranial and upper torso anatomy relative to first image taken
Change in number of detectable anatomical landmarks after patient residual motion | 20 minutes
  Change in number of detection of points in the point cloud in response to residual motion of anatomical landmarks over 20 minutes of continuous data acquisition
Photograph record of physical characteristics of face and hair that may affect detection of anatomical landmarks by the surface monitoring system | 5 seconds
  A photograph taken by the system camera showing physical characteristics of face and hair (e.g. shape, tone, location, size)
Effect of change in participants' weight (kg) from pre_RT to late RT on absolute residual motion of cranial and upper torso anatomy | 4 to 6 weeks
  The effect of change in weight (kg) from pre-RT to late RT on Outcome 5
Effect of change in participants' weight (kg) from pre_RT to late RT on relative residual motion of cranial and upper torso anatomy | 4 to 6 weeks
  The effect of change in weight (kg) from pre-RT to late RT on Outcome 6

CONTACTS AND LOCATIONS:
Overall Officials: Purmina Sundaresan, Dr, Principal Investigator — Western Sydney Local Health District
Locations (1):
- Blacktown Hospital, Blacktown, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Non-identifiable individual participant data (IPD) may be shared with researchers for further scientific research. Facial images/photos identifying participants will not be shared.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Not before the study completion. For not more than 15 years after study completion, at which time the data sharing plan will be revised.